CLINICAL TRIAL: NCT03658473
Title: Double-blind, Phase III Study to Evaluate Gastroprotection Obtained by the Use of Rebamipide 300 mg (2x Daily) and Rabeprazole 20 mg/Day (1x Daily) Associated or Not to Prevent Naproxen (1100 mg/Day)-Induced Gastric Lesions for 7 Days.
Brief Title: Evaluation of Rebamipide and Rabeprazole Effect Associated or Not to Prevent Naproxen-induced Gastric Lesions
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Galeno Desenvolvimento de Pesquisas Clínicas (Other Government)
Collaborators: Biolab Sanus Farmaceutica (Industry)
Responsible Party: Principal Investigator, Gilberto De Nucci, Doctor, Galeno Desenvolvimento de Pesquisas Clínicas
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: GDN 005/15
Record Dates: First submitted 2018-09-01; First posted 2018-09-05 (Actual); Last update posted 2018-09-05 (Actual); Status verified 2018-09

CONDITIONS: Gastric Lesion
Keywords: gastroprotection; rebamipide; rabeprazole; naproxeno
MeSH Terms: interventions — Naproxen; rebamipide; Rabeprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Treatment A (Active Comparator): Administration of 550 mg naproxen 2x daily + 300 mg rebamipide 2x daily + 20 mg rabeprazole 1x daily over 7 days.
  Interventions: Drug: 550 mg naproxen + 300 mg rebamipide + 20 mg rabeprazole.
- Treatment B (Active Comparator): Administration of 550 mg naproxen 2x daily + 300 mg rebamipide placebo 2x daily + 20 mg rabeprazole 1x daily over 7 days.
  Interventions: Drug: 550 mg naproxen + placebo + 20 mg rabeprazole
- Treatment C (Active Comparator): Administration of 550 mg naproxen 2x daily + 300 mg rebamipide 2x daily + 20 mg rabeprazole placebo 1x daily over 7 days.
  Interventions: Drug: 550 mg naproxen + 300 mg rebamipide + placebo
- Treatment D (Placebo Comparator): Administration of 550 mg naproxen 2x daily + 300 mg rebamipide placebo 2x daily + 20 mg rabeprazole placebo 1x daily over 7 days.
  Interventions: Drug: 550 mg naproxen + placebo + placebo

INTERVENTIONS:
Drug: 550 mg naproxen + 300 mg rebamipide + 20 mg rabeprazole. — Oral administration of 550 mg naproxen 2x daily + 300 mg rebamipide 2x daily + 20 mg rabeprazole 1x daily over 7 days.
  Arms: Treatment A
Drug: 550 mg naproxen + placebo + 20 mg rabeprazole — Oral administration of 550 mg naproxen 2x daily + placebo of rebamipide 2x daily + 20 mg rabeprazole 1x daily over 7 days.
  Arms: Treatment B
Drug: 550 mg naproxen + 300 mg rebamipide + placebo — Oral administration of 550 mg naproxen 2x daily + 300 mg rebamipide 2x daily + placebo of rabeprazole 1x daily over 7 days.
  Arms: Treatment C
Drug: 550 mg naproxen + placebo + placebo — Oral administration of 550 mg naproxen 2x daily + placebo 2x daily + placebo of rabeprazole 1x daily over 7 days.
  Arms: Treatment D

SUMMARY:
This clinical trial evaluated the gastroprotection obtained by the use of rebamipide 300 mg (2x daily) and rabeprazole 20 mg/day (1x daily) associated or not in the prevention of gastric lesions induced by naproxen 1100 mg/day) for 7 days to healthy volunteers of both sexes. This trial also assessed drugs safety and tolerability, the prostaglandin levels (PGE2) in biopsy specimens before and after treatment of each group and the histopathological changes induced by the treatment of each group.

DETAILED DESCRIPTION:
This phase III, single center, double-blind, randomised, multiple-dose trial was performed in a parallel-group design. The subjects were randomly assigned to one of the 4 possible treatments: treatment A - 550 mg naproxen 2x daily + 300 mg rebamipide 2x daily + 20 mg rabeprazole 1x daily over 7 days; treatment B - 550 mg naproxen 2x daily + placebo of rebamipide 2x daily + 20 mg rabeprazole 1x daily over 7 days; treatment C - 550 mg naproxen 2x daily + 300 mg rebamipide 2x daily + placebo of rabeprazole 1x daily over 7 days; and treatment D - 550 mg naproxen 2x daily + placebo of rebamipide 2x daily + placebo of rabeprazole 1x daily over 7 days.

Upper digestive endoscopy was performed before the beginning of the therapies and 12 hours after the last administration (8th day of the study), with collection of the biological samples (biopsies) in the antrum region and 5 in the gastric body at each examination. The samples were preserved in formalin solution and sent for histopathological examination.

The safety and tolerability was assessed by signs and symptoms, adverse events, laboratory tests, vital signs and electrocardiogram (ECG).

ELIGIBILITY:
Inclusion Criteria:

* Volunteers of both sexes aged 18 or over. Women could not be pregnant or breastfeeding
* Body-mass index (BMI) ≥19.0 kg/m² and ≤ 28.75 kg/m²
* Good state of health
* Non-smoker or ex-smoker for at least 6 month
* Written informed consent, after having been informed about benefits and potential risks of the clinical trial, as well as details of the insurance taken out to cover the subjects participating in the clinical trial

Exclusion Criteria:

* Existing cardiac, hepatic and/or haematological diseases or pathological findings, which might interfere with the safety or tolerability and/or pharmacokinetics and/or pharmacodynamics of the active ingredient
* History of relevant central nervous system (CNS) and/or psychiatric disorders and/or currently treated CNS and/or psychiatric disorders
* Known allergic reactions to the active ingredients used or to constituents of the pharmaceutical preparations
* Subjects with severe allergies or multiple drug allergies, unless it is judged as not relevant for the clinical trial by the investigator
* Volunteer does not present the entire upper gastrointestinal tract mucosa, that is, hemorrhages, ulcers or apparent lesions at the first endoscopic examination.
* The volunteer that has achlorhydria (intragastric pH greater than 6.5)
* Occult blood in the faeces with positive result before the start of therapy
* Electrocardiographic findings not recommended by the researcher for participation in the study
* Deviations from the results of laboratory recruitment examinations considered clinically relevant by the researcher
* Has a history of alcohol or drug abuse or expressive alcohol consumption (> 35g/day)
* Participation in a clinical trial during the last 6 months prior to individual enrolment of the subject
* Have used regular medication within 2 weeks prior to initiation of treatment or used any medication within one week prior to initiation of study treatment, with the exception of oral contraceptives or cases where, based on half-life of the drug and/or active metabolites, complete elimination may be assumed
* Subjects who are unable to understand the written and verbal instructions, in particular regarding the risks and inconveniences they will be exposed to during their participation in the clinical trial

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2014-11-12 (Actual); Primary Completion 2014-11-27 (Actual); Study Completion 2015-02-04 (Actual)

PRIMARY OUTCOMES:
Evaluation of the number of gastric events (erosion of the gastric mucosa, gastritis, petechiae in the gastric mucosa and ulcer) | 0-7 days after drugs administration
  Histopathological examination of biological samples (biopsies) in the antrum region and in the gastric body collected during the upper digestive endoscopy performed before the beginning of the therapies and 12 hours after the last administration (8th day of the study) to each subject.

SECONDARY OUTCOMES:
Measurement of prostaglandin levels (PGE2). | 0-7 days after drugs administration
  Measurement of prostaglandin levels (PGE2) in biopsy specimens collected before and after treatment of each subject.
Number of adverse events per participant | 0-7 days after drugs administration
  Number of adverse events in each treatment group, including clinically relevant alterations of vital signs and laboratory tests results.

CONTACTS AND LOCATIONS:
Overall Officials: Gilberto De Nucci, Doctor, Principal Investigator — Galeno Desenvolvimento de Pesquisas Clinicas Ltda
Locations (1):
- Galeno Desenvolvimento de Pesquisas Clinicas Ltda., Campinas, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No